CLINICAL TRIAL: NCT04936828
Title: Ecological Momentary Intervention for Stroke Caregivers' Psychological Support: a Randomised Controlled Trial
Brief Title: Ecological Momentary Intervention for Stroke Caregivers' Psychological Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17617620
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Caregiver Burnout; Depressive Symptoms; Psychological Distress; Mobile Phone Use
MeSH Terms: conditions — Stroke; Caregiver Burden; Depression; Cell Phone Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receive iCBT based EMI with message content, delivery frequency and timing personalised to participants' preferences.
  Interventions: Other: iCBT-based EMI
- Control group (No Intervention): Receive general mental health information through instant message.

INTERVENTIONS:
Other: iCBT-based EMI — Consists of brief iCBT for psychological support (mandatory), stroke care education (optional), and nurse-led real-time chat-based support messages, delivered according to participants' preferences.
  Arms: Intervention group

SUMMARY:
The proposed trial aims to evaluate the effectiveness of internet-delivered cognitive behavioural therapy (iCBT) based ecological momentary intervention (EMI) for psychological well-being in stroke family caregivers.

DETAILED DESCRIPTION:
Many stroke patients require long-term care in the community. In Hong Kong (HK), most stroke caregivers in the community are family members, and many require psychological support for caregiver stress. However, these caregivers have difficulties accessing existing centre-based services due to varying work and care responsibilities, and therefore require alternative support services to meet their unique needs and schedules. Evidence shows that internet-delivered cognitive behavioural therapy (iCBT) is effective in managing psychological distress including depressive symptoms, especially when guided by healthcare professionals. Ecological momentary intervention (EMI) is an innovative and cost-effective intervention 'framework' that utilises mobile messages to deliver personalised psychological interventions. The proposed trial aims to deliver iCBT-based EMI through instant messaging applications (e.g. WhatsApp) to provide personalised and real-time psychological support led by nurses. Screened stroke caregivers with Patient Health Questionnaire-9 (PHQ-9) scores ranging from 5 to 19 (mild to moderately severe depressive symptoms) will be recruited from community centres, rehabilitation centres and outpatient clinics in HK. They will then be individually randomised into the Intervention group (n=128) or Control group (n=128). The Intervention group will receive the iCBT-based EMI for 12 weeks, which includes instant messages sent at the times and frequencies of the participants' choosing, and chat-based psychological support led by nurses to enhance effects of iCBT through real-time counselling and practical advice. The control group will only receive instant messages on general mental health information and reminders to participate in follow-up surveys. The primary outcome is PHQ-9 scores at 24 weeks. Secondary outcomes will include anxiety, perceived stress, caregiver burden, caring experience, spiritual well-being and quality-of-daily-life. We will strictly follow the CONSORT-EHEALTH checklist. A post-trial qualitative study will be conducted to understand the participants' experience of and compliance with the EMI. The intervention will be highly applicable for all caregivers requiring psychological support and will be one step further in meeting the World Health Organization's recommendations in supporting caregivers in the context of global ageing populations.

ELIGIBILITY:
Inclusion Criteria:

* Primary family caregiver of stroke patient (modified Barthel Index [mBI] <15; usually represent moderate disability)
* Able to read and communicate in Chinese
* Aged ≥18
* Able to use mobile phone text messaging function
* PHQ-9 ranged from 5 to 19

Exclusion Criteria:

* Professional medical personnel and professional carer
* Has provided care for <1 month prior to recruitment
* Has diagnosis of psychiatric disease or is currently taking psychotropic drug
* PHQ-9 ≥ 20 (i.e., severe depressive symptom)
* Currently participating in any type of psychological intervention (e.g., CBT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms (Patient Health Questionnaire-9 [PHQ-9]) | 24-week
  A 9-item scale with score ranging from 0 to 27, higher scores indicate higher severity of depressive symptom

SECONDARY OUTCOMES:
Anxiety symptoms (Generalized Anxiety Disorder-7 [GAD-7]) | 24-week
  A 7-item scale with score ranging from 0 to 21, higher scores indicate higher severity of anxiety symptoms
Stress level (Perceived Stress Scale [PSS-4]) | 24-week
  A 4-item scale with score ranging from 0 to 16, higher scores indicate higher severity of stress
Caregiver's burden (Zarit Burden Interview [ZBI-4]) | 24-week
  A 4-item scale with score ranging from 0 to 16, higher scores indicate higher severity of caregiving burden
Caring experience (Positive Aspects of Caregiving [PAC]) | 24-week
  An 11-item scale with score ranging from 0 to 44, higher scores indicate more positive appraisal of caregiving experience
Spiritual well-being (Sub-scale of Spirituality Scale for Chinese Elders [SSCE]) | 24-week
  An 8-item scale with score ranging from 0 to 32, higher scores indicate better spiritual well-being
Quality of life (EuroQol 5-dimension 5-level questionnaire [EQ-5D-5L]) | 24-week
  A 5-item scale with predicted values ranging from -.864 to 1, higher values indicate higher health-related quality of life

CONTACTS AND LOCATIONS:
Locations (7):
- Hong Kong (7):
  - Hong Kong PHAB Association, Hong Kong
  - Hong Kong Stroke Association, Hong Kong
  - NT West Community Rehabilitation Day Centre, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Hong Kong Society for Rehabilitation, Hong Kong
  - Tung Wah Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No